CLINICAL TRIAL: NCT05114629
Title: Biomechanics of Adaptive Rowing in Active and Inactive Manual Wheelchair Users
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 20-01368
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Wheelchair; Water Sports; Upper Extremity; Biomechanics; Electromyography; Kinematics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Individuals in the active group will meet or exceed the American College of Sports Medicine's Guidelines for Physical Activity in Adults with Chronic Health Conditions and Disabilities. ACMS recommends individuals participate in at least 150 to 300 minutes of moderate-intensity aerobic exercise, 75 to 150 minutes of vigorous-intensity activity.(health.gov/ PAGuidelines)
- Inactive: Individuals in the inactive group are those who do not meet the American College of Sports Medicine's Guidelines for Physical Activity in Adults with Chronic Health Conditions and Disabilities. ACMS recommends individuals participate in at least 150 to 300 minutes of moderate-intensity aerobic exercise, 75 to 150 minutes of vigorous-intensity activity.(health.gov/ PAGuidelines)

SUMMARY:
This research is being performed to characterize the rowing stroke in active and inactive individuals who use a manual wheelchair. The investigators will be looking at muscle activity of four shoulder muscles (upper trapezius, lower trapezius, serratus anterior, and posterior deltoid) and motion of the arms, shoulder blade, and trunk during rowing. This will be done for three rowing conditions (1: adapted rowing ergometer, 2: rowing ergometer from a chair, 3: standard seated row exercise using an elastic band [TheraBand]). The investigators are also looking at shoulder strength, range of motion, quality of life, and community participation.

DETAILED DESCRIPTION:
Individuals who use a manual wheelchair (MWC) are at a high risk of developing long-term shoulder pain and impairment caused by increased demand and load on the shoulder during normal daily activities. Two main contributors to shoulder pain are overuse and shoulder muscle imbalance. Rehabilitation programs targeting shoulder pain suggest stretching anterior shoulder muscles and strengthening posterior shoulder muscles to promote balance and stability across the shoulder. Rowing-type exercises have been shown to be beneficial in accomplishing this. In addition to reducing shoulder pain, it is crucial to identify methods and modes of exercise which are more widely accessible. Participation in physical activity provides physical, psychological, and social benefits. However, several barriers to physical activity have been reported in this population. Less than half of individuals with physical disabilities meet the American College of Sports Medicine's physical activity guidelines.

The primary aim of this study is to determine the biomechanics of the rowing stroke in active and inactive individuals who use a MWC for mobility. Muscle activity (electromyography) of four shoulder muscles (upper trapezius, lower trapezius, serratus anterior, and posterior deltoid) and 3D motion analysis of the arms, shoulder blade, and trunk will be analyzed across three rowing conditions (adapted rowing ergometer, rowing ergometer from chair, standard row exercise). The investigators hypothesize rowing on the adapted rowing ergometer will lead to greater muscle activity than the standard rowing exercise and there will be no difference in arm, shoulder blade, and trunk movement between rowing conditions. The secondary aim of this study is to assess shoulder range of motion, pectoralis minor muscle extensibility, quality of life, and community participation. The investigators hypothesize active individuals will have a greater range of motion and pectoralis minor muscle extensibility and report lower quality of life and community participation than inactive individuals. This study seeks to lay the groundwork of evidence to suggest participation in rowing as a viable option to reduce the frequency and intensity of shoulder pain and provide a more accessible form of physical activity. Additionally, the investigators hope to contribute further insight into clinical measures (shoulder strength, range of motion, pectoralis minor muscle extensibility), subjective quality of life, and community participation in this population.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years of age
* use a manual wheelchair for at least 50% of community mobility
* able to transfer independently (with or without the use of adaptive equipment)
* able to achieve humeral elevation of greater than or equal to 90 degrees (bilaterally)
* cleared for exercise participation as indicated by the ACSM Preparticipation Health Screening (Riebe et al., 2015)
* able to read and understand English

Exclusion Criteria:

* have an active pressure sore or skin breakdown
* have a presence of shoulder pain as indicated by a score of greater than 12 on the Wheelchair Users Shoulder Pain Index (Mulroy et al., 2015)
* have impaired upper extremity function as indicated by a score of greater than 40 on the QuickDASH (Angst et al., 2011; Kennedy et al., 2011)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited through personal contact, using flyers, newsletters, email communication, and social media. Participants will be recruited from the community in the Greater Philadelphia area through previously established connections at the Philadelphia Center for Adapted Sports (PCAS) and Magee Rehabilitation Network, as well as through social media platforms (Facebook, Instagram) and the Drexel University College of Nursing and Health Professions webpage.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Electromyography | Collected during Day 2 visit
  Surface EMG will be used to determine levels of muscle activation through analyzing area under the curve, peak, and mean amplitude. Data will be collected on four muscles bilaterally (upper trapezius, lower trapezius, serratus anterior, and posterior deltoid).Peak dynamic method will be used for normalization for comparison between exercise conditions.(Ryan et al., 1992; Fleming & Donne, 2014; Hug & Dorel, 2009)
Kinematics | Collected during Day 2 visit
  Three-dimensional kinematic data of the trunk, arms, and scapula will be collected using the Motion Monitor electromagnetic transmitter system (Innovative Sports Training, Inc., Chicago, IL). The International Society of Biomechanics recommendations for shoulder kinematics, will be used to define sensor placement and global and local coordinate system definitions.(Wu et al., 2005) Using this data, we will analyze the coordination and symmetry of the upper extremity during the rowing stroke to supplement the EMG data.

SECONDARY OUTCOMES:
Shoulder Muscle Strength | Collected during Day 1 visit
  Shoulder girdle strength will be measured bilaterally using a handheld dynamometer (HHD) (Lafayette Manual Muscle Tester, Lafayette, IN). Flexion, extension, abduction, adduction, internal, and external rotation strength will be measured. Standard manual muscle testing positions, as previously described by Kendall et al., 2005 will be used with a modification to allow participants to remain in their wheelchairs during testing. Peak force, measured in kilograms (kg), will be normalized to body weight (BW) for comparison across participants [%BW=(forcekg/BWkg)*100].
Shoulder Range of Motion | Collected during Day 1 visit
  Active shoulder ROM will be measured bilaterally for elevation, extension, external rotation (humerus in 90° elevation), and internal rotation. ROM will be measured using goniometer and analyzed using the maximum value recorded over two trials.
Subjective quality of life | Collected During Day 1 visit
  The SQoL is a self-report questionnaire measuring the individual's overall perception of their quality of life. The SQoL consists of one question asking individuals to rate their overall quality of life taking everything into account. The question is measured using a Likert-type scale where 1 = life is very distressing, it's hard to imagine how it could get much worse; to 7 = life is great, it's hard to imagine how it could get much better.(Dijkers, 2005)
Community Participation | Collected during Day 1 visit
  The Community Participation Indicators' Enfranchisement Scale (CPI) will be used to measure community participation. The CPI is a 48-question self-report questionnaire measuring two domains of community participation, importance of participation and control over participation.(Heinemann et al., 2013) Questions are answered by selecting one of five options: "all the time, frequently, sometimes, seldom, and almost never". The score is broken down by domain and scores range from 0 to 100 for each domain. A higher score is indicative of greater participation.
Descriptive Variables | Collected during Day 1 visit
  Descriptive variables will be collected including age, gender, race, ethnicity, education, socioeconomic status, self-reported general medical history and history of health condition/injury; wheelchair specifics.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Euiler, MS, Principal Investigator — Drexel University
Locations (1):
- Elizabeth Euiler, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided